CLINICAL TRIAL: NCT02414880
Title: Sugammadex Versus Neostigmine for Antagonism of Rocuronium-induced Neuromuscular Blockade in Patients With Liver Cirrhosis Undergoing Liver Resection: A Controlled Randomized Study
Brief Title: Sugammadex Versus Neostigmine in Patients With Liver Cirrhosis Undergoing Liver Resection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: National Liver Institute, Egypt (Other)
Responsible Party: Principal Investigator, Professor Mohamed Abdulatif Mohamed, Prof. Mohamed Abdulatif Mohamed, MD, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Suga-Neo
Record Dates: First submitted 2015-04-05; First posted 2015-04-13 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Cirrhosis and Chronic Liver Disease
Keywords: Sugammadex; Neostigmine; Rocuronium; Cirrhosis; Liver resection; Neuromuscular
MeSH Terms: conditions — Fibrosis | interventions — Sugammadex; Neostigmine; Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sugammadex/ Normal liver (Active Comparator): Patients with American Society of Anesthesiologists physical status (ASA) class I with normal preoperative liver functions undergoing liver resection.
  Rocuronium-induced neuromuscular blockade will be reversed at the end of the operation when two responses to train-of-four ulnar nerve stimulation are detected (T2) by injection of sugammadex 2mg/kg.
  Interventions: Drug: Sugammadex; Drug: Rocuronium
- Neostigmine / Normal liver (Active Comparator): Patients with American Society of Anesthesiologists physical status (ASA) class I with normal preoperative liver functions undergoing liver resection.
  Rocuronium-induced neuromuscular blockade will be reversed at the end of the operation when two responses to train-of-four ulnar nerve stimulation are detected (T2) by injection of neostigmine 50 micro-gram/kg combined with atropine 20 micro-gram/kg.
  Interventions: Drug: Neostigmine; Drug: Rocuronium
- Sugammadex / Liver cirrhosis (Active Comparator): Patients with liver cirrhosis, Child classification "A" with a Model for End-Stage Liver Disease (MELD) score <10 undergoing liver resection.
  Rocuronium-induced neuromuscular blockade will be reversed at the end of the operation when two responses to train-of-four ulnar nerve stimulation are detected (T2) by injection of sugammadex 2mg/kg.
  Interventions: Drug: Sugammadex; Drug: Rocuronium
- Neostigmine / Liver cirrhosis (Active Comparator): Patients with liver cirrhosis, Child classification "A" with a Model for End-Stage Liver Disease (MELD) score <10 undergoing liver resection.
  Rocuronium-induced neuromuscular blockade will be reversed at the end of the operation when two responses to train-of-four ulnar nerve stimulation are detected (T2) by injection of neostigmine 50 micro-gram/kg combined with atropine 20 micro-gram/kg.
  Interventions: Drug: Neostigmine; Drug: Rocuronium

INTERVENTIONS:
Drug: Sugammadex — Rocuronium-induced neuromuscular blockade will be reversed at the end of the operation when two responses to train-of-four ulnar nerve stimulation are detected (T2) by injection of sugammadex 2mg/kg.
  Other Names: Bridion
  Arms: Sugammadex / Liver cirrhosis; Sugammadex/ Normal liver
Drug: Neostigmine — Rocuronium-induced neuromuscular blockade will be reversed at the end of the operation when two responses to train-of-four ulnar nerve stimulation are detected (T2) by injection of neostigmine 50 micro-gram/kg combined with atropine 20 micro-gram/kg.
  Other Names: Prostigmine
  Arms: Neostigmine / Liver cirrhosis; Neostigmine / Normal liver
Drug: Rocuronium — An intubating dose of Rocuronium (0.6 mg/kg) will be given with induction of anesthesia and the degree of muscle relaxation will be evaluated through out the operation by recording the response of the hand muscles to train-of-four ulnar nerve stimulator (Mechanosensor Neuromuscular Transmission Module of General Electric AISYS Anaesthesia machine USA) according to the Good Clinical Research Practice (GCRP) guidelines for pharmacodynamic neuromuscular studies. Muscle relaxation will be maintained by additional top-up doses of Rocuronium (0.15mg/kg) which will be administered after detection of the first response to TOF stimulation (T1).
  Other Names: Esmeron

SUMMARY:
Liver cirrhosis is a progressive disease characterized by loss of functional hepatocytes that substantially affects drug pharmacokinetics. Rocuronium onset time is longer and recovery time from it is prolonged in cirrhotic patients than in those with normal liver function.

This randomized controlled study is designed to compare the pharmacodynamic profiles of sugammadex and neostigmine when used for the antagonism of moderate degree of rocuronium-induced neuromuscular block in cirrhotic patients undergoing liver resection and in patients with preoperative normal liver functions undergoing liver resection.

DETAILED DESCRIPTION:
Liver resection is a lengthy operation that has major effects on patient hemodynamics and perioperative liver functions. These effects are more obvious in patients with liver cirrhosis. Liver cirrhosis is a progressive disease characterized by loss of functional hepatocytes that substantially affects drug pharmacokinetics.

Rocuronium is an intermediate acting steroidal non-depolarizing neuromuscular blocker that is mostly metabolized by the liver. Its onset time is longer in cirrhotic patients than in those with normal liver function. This can be explained by an increase in the volume in which it initially distributes. Although elimination kinetics are unchanged in patients with cirrhosis, Rocuronium recovery time is prolonged in cirrhotic patients.

To speed up the process of antagonism of residual neuromuscular blockade, inhibitors of acetyl cholinesterases such as Neostigmine are usually administered only when there is evidence of spontaneous recovery of neuromuscular function. Too early administration of Neostigmine is not effective and may produce serious side-effects from accumulation of Acetylcholine in other organs, especially the brain and heart.

Sugammadex, a modified γ-cyclodextrin, is the first selective relaxant binding agent. It forms very tight, stable complexes in a 1:1 ratio with Rocuronium. The inactive Sugammadex-Rocuronium complex undergoes renal elimination. Sugammadex has no effect on acetyl cholinesterases or on any receptor system in the body, eliminating the need for anticholinergic drugs. Sugammadex can antagonize any level of neuromuscular blockade, including the profound blockade induced by Rocuronium.

The use of Sugammadex in different patient populations including end-stage renal failure is associated with consistent, complete and rapid recovery of neuromuscular functions. It is of clinical relevance to note that in the presence of Sugammadex, the hepatic biotransformation and final clearance of Rocuronium via biliary excretion is changed to a completely different (liver-independent) renal pathway. A recent report described the successful use of Sugammadex to antagonize prolonged deep rocuronium-induced neuromuscular block in patients with normal liver functions undergoing liver resection. Furthermore, the successful use of Sugammadex to antagonize Rocuronium neuromuscular block was also reported in a case series of three patients with liver dysfunction.

To the best of our knowledge, there are no controlled randomized studies evaluating the use of Sugammadex to antagonize residual Rocuronium-induced neuromuscular blockade in patients with liver cirrhosis undergoing open surgical liver resection. This randomized controlled study is designed to compare the pharmacodynamic profiles of Sugammadex and Neostigmine when used for the antagonism of moderate degree of Rocuronium-induced neuromuscular block in cirrhotic patients undergoing liver resection and in patients with preoperative normal liver functions undergoing liver resection.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status (ASA) class I for patients with preoperative normal liver function test (two groups) and I-III for patients with liver cirrhosis (two groups).
* For the two "Liver Cirrhosis" groups: Patients with liver Cirrhosis with Child classification "A" and a Model for End-Stage Liver Disease (MELD) score <10 undergoing Liver resection surgeries.
* For the two "Normal Liver" groups: Patients with normal preoperative liver functions undergoing Liver resection surgeries.

Exclusion Criteria:

* Co-existing neuromuscular disease.
* Body mass index more than 35 kg/m-2.
* Renal impairment.
* Medications known to affect neuromuscular transmission (e.g. Aminoglycoside antibiotics or Magnesium Sulphate).
* Bleeding tendency.
* Intra-operative adverse events (e.g. massive bleeding or hypothermia).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The time from reversal to Train-of-four (TOF) ratio of 0.9 | 15 min
  The time from the administration of Sugammadex or Neostigmine till recovery of the TOF ratio to 0.9

SECONDARY OUTCOMES:
The time from reversal to Train-of-four (TOF) ratio of 1 | 30 min
  The time from the administration of Sugammadex or Neostigmine till recovery of the TOF ratio to 1.
Length of stay in the post-anesthesia care unit (PACU) | 4 hours
  Time required in post-anesthesia care unit (PACU) to achieve a modified Aldrete score of 9
Time from last Rocuronium dose to Train-of-four (TOF) ratio of 0.9 | 1 hour
  The time from the last dose of Rocuronium to recovery of the TOF ratio to 0.9.
Duration of action of the initial intubating dose of Rocuronium | 45 min
  The time interval between the initial Rocuronium intubating dose administration and the recovery of the first twitch of the TOF response (T1).
Incidence of postoperative re-curarization | 4 hours
  Recurrence of neuromuscular block (re-curarization) will be defined as a decrease in the TOF ratio to <0.9 after full recovery had been detected, or as a deterioration in the clinical signs of recovery from the block.
Total dose of Rocuronium | 24 hours
  Total dose of Rocuronium used during the whole operation including the intubating dose and the subsequent top-ups.
Duration of anesthesia | 24 hours
  Duration between induction of anesthesia and complete recovery of consciousness and motor power.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdulatif Mohamed, M.D., Principal Investigator — Cairo University
Locations (1):
- National Liver institute, Ḩadā’iq al Qubbah, Cairo Governorate, Egypt

REFERENCES:
- [Background] Schaller SJ, Fink H. Sugammadex as a reversal agent for neuromuscular block: an evidence-based review. Core Evid. 2013;8:57-67. doi: 10.2147/CE.S35675. Epub 2013 Sep 25. PMID 24098155
- [Background] Edginton AN, Willmann S. Physiology-based simulations of a pathological condition: prediction of pharmacokinetics in patients with liver cirrhosis. Clin Pharmacokinet. 2008;47(11):743-52. doi: 10.2165/00003088-200847110-00005. PMID 18840029
- [Background] Kopman AF, Eikermann M. Antagonism of non-depolarising neuromuscular block: current practice. Anaesthesia. 2009 Mar;64 Suppl 1:22-30. doi: 10.1111/j.1365-2044.2008.05867.x. PMID 19222428
- [Background] Caldwell JE. Clinical limitations of acetylcholinesterase antagonists. J Crit Care. 2009 Mar;24(1):21-8. doi: 10.1016/j.jcrc.2008.08.003. Epub 2009 Jan 17. PMID 19272535
- [Background] Naguib M. Sugammadex: another milestone in clinical neuromuscular pharmacology. Anesth Analg. 2007 Mar;104(3):575-81. doi: 10.1213/01.ane.0000244594.63318.fc. PMID 17312211
- [Background] Nonaka T, Fujimoto M, Nishi M, Yamamoto T. [The effect of rocuronium and sugammadex in hepatic tumor patients without preoperative hepatic impairment]. Masui. 2013 Mar;62(3):304-8. Japanese. PMID 23544332
- [Background] Batistaki C, Matsota P, Kalimeris K, Brountzos E, Kostopanagiotou G. Sugammadex antagonising rocuronium in three patients with liver dysfunction undergoing transjugular intrahepatic portosystemic shunt. Anaesth Intensive Care. 2012 May;40(3):556-7. No abstract available. PMID 22577926
- [Background] Blobner M, Eriksson LI, Scholz J, Motsch J, Della Rocca G, Prins ME. Reversal of rocuronium-induced neuromuscular blockade with sugammadex compared with neostigmine during sevoflurane anaesthesia: results of a randomised, controlled trial. Eur J Anaesthesiol. 2010 Oct;27(10):874-81. doi: 10.1097/EJA.0b013e32833d56b7. PMID 20683334
- [Background] Illman HL, Laurila P, Antila H, Meretoja OA, Alahuhta S, Olkkola KT. The duration of residual neuromuscular block after administration of neostigmine or sugammadex at two visible twitches during train-of-four monitoring. Anesth Analg. 2011 Jan;112(1):63-8. doi: 10.1213/ANE.0b013e3181fdf889. Epub 2010 Oct 26. PMID 20978247